CLINICAL TRIAL: NCT00404950
Title: Effects of Hyperglycemia During Cardiopulmonary Bypass on Renal Function
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0408007400
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Hyperglycemia; Diabetes
Keywords: hyperglycemia; cardiopulmonary bypass; renal injury; diabetes
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — At the following times when plasma glucose will be measured, an additional 6 mL of blood will be drawn (from indwelling routine arterial line catheter) into EDTA tubes and immediately centrifuged: baseline following induction, once during cardiopulmonary bypass, at arrival in the intensive care unit, and the morning after surgery- totaling 24 mls of blood. The platelet rich plasma will be withdrawn and one half of the volume immediately frozen for subsequent HPLC measurement of BH2 and BH4. The remaining plasma will be subjected to progressive centrifugation steps in order to concentrate the platelet fraction that will then be suspended in buffer and frozen. VASP expression and phosphorylation will be determined by Western blot.
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine whether intraoperative hyperglycemia potentiates renal injury in the setting of cardiac surgery requiring cardiopulmonary bypass.

DETAILED DESCRIPTION:
Significance:

Postoperative renal dysfunction is a common complication of cardiopulmonary bypass occurring in nearly 8% of all patients undergoing myocardial revascularization. Both diabetes and preoperative hyperglycemia are independent risk factors for postoperative renal dysfunction after coronary artery bypass surgery.

The cause of renal injury is multifactoral and in most cases involves renal ischemia from alteration of renal perfusion, resistance, metabolic byproducts (free-radical species), inflammatory mediators and embolic processes.

In the setting of ischemia, specifically, neuronal, hyperglycemia has been shown to worsen neurologic outcome and interfere with wound healing-possibly increasing the incidence of wound infection.

Hyperglycemia is common during cardiopulmonary bypass in both diabetic and non-diabetic patients as a result of altered glucose regulation during hypothermic conditions (body temperature actively cooled to 28 degree centigrade) and, more importantly, from delivery of cardioplegia to arrest the heart allowing for surgical repair in a non-beating heart. The cardioplegia is rich in potassium, among other agents, believed to offer cardioprotection during cardiopulmonary bypass and is prepared in Dextrose 5% and normal saline. On average, each patient receives nearly 2 liters of this solution, amounting to 100 grams or more of glucose. In this setting, hyperglycemia is also promoted from insulin suppression, stress hormone induced gluconeogenesis and enhanced tubular resorption.

Only recently have perioperative clinicians become aware about potential ischemic effects of hyperglycemia during bypass and the need to maintain 'tight' control of glucose to avoid stroke. This practice, however, is inconsistent and mostly applied to diabetic patients.

We hypothesize that tubular injury may be exacerbated by hyperglycemia in non-diabetic patients while undergoing hypothermic cardiopulmonary bypass and have undertaken this prospective observational study to investigate the relationship between intraoperative glucose and postoperative renal dysfunction.

Methodology:

We plan to study to 200 patients ≥ 50 years of age scheduled for procedures requiring cardiopulmonary bypass whether for coronary revascularization or valvular surgery. After informed consent is obtained each patient's preoperative lab values consisting of serum glucose, urine glucose, creatinine and BUN will be noted. Each patient's pre-induction hemodynamics will also be noted. During bypass, serum and urine glucose will be measured every 20 minutes in addition to collecting information on temperature of cardioplegic solution, lowest patient temperature, time of bypass, and use of diuretics, or vasoactive drugs. Additional sampling of serum creatinine and glucose and vital signs will take place upon arrival in the cardiac intensive care unit after surgery and throughout hospitalization as is standard of care in cardiac surgery at this institution. No extra samples will be taken but the standard measurements will be observed. The clinical outcome of interest is a new onset of renal dysfunction defined as a post-operative serum creatinine change of 0.5 mg/dl or greater after surgery.

Inclusion Criteria:

1. Male and female patients ≥ 50 years of age
2. Patients undergoing on pump cardiopulmonary bypass for either myocardial revascularization (coronary artery bypass graft) or valvular surgery (valve repair or replacement)

Exclusion Criteria:

1. Patients with insulin dependent diabetes
2. Patients with preexisting renal dysfunction defined as Creatinine> 2 mg/dl
3. Patients in need of emergency cardiac procedures

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥ 50 years of age
2. Patients undergoing on pump cardiopulmonary bypass for either myocardial revascularization (coronary artery bypass graft) or valvular surgery (valve repair or replacement)

Exclusion Criteria:

1. Patients with insulin dependent diabetes
2. Patients with preexisting renal dysfunction defined as Creatinine> 2 mg/dl
3. Patients in need of emergency cardiac procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing on pump cardiopulmonary bypass for either myocardial revascularization (coronary artery bypass graft) or valvular surgery (valve repair or replacement)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2005-07 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Heerdt, MD, PhD, Principal Investigator — Associate Professor
Locations (1):
- The New York Presbyterian Hospital - Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Will not share